CLINICAL TRIAL: NCT05953831
Title: Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Safety and Efficacy Study of CDR132L on Reverse Cardiac Remodeling in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction and Cardiac Hypertrophy
Brief Title: Reverse Remodeling Effects of CDR132L in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction and Cardiac Hypertrophy
Acronym: REMOD-REVERT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Transfer of study responsibility and planning
Sponsor: Cardior Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR132L-P2-06
Record Dates: First submitted 2023-06-29; First posted 2023-07-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF; Heart failure; Cardiac Hypertrophy
MeSH Terms: conditions — Heart Failure; Cardiomegaly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IMP to be masked after preparation by unblinded staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CDR132L 4.52 mg (Experimental): Six times CDR132L 4.52 mg/kg body weight intravenous in single dose.
  Interventions: Drug: CDR132L
- Placebo (Placebo Comparator): Six times Placebo intravenous in single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CDR132L — CDR132L is a synthetic antisense oligonucleotide (ASO) and a selective inhibitor of microRNA-132-3p (miR-132). miR-132 in cardiomyocytes is a central switch affecting the expression of genes that are crucially involved in maladaptive cardiac remodeling, transformation, and pathological cardiac growth (hypertrophy), contributing to adverse cardiac remodeling and heart failure (HF).1-5 Aberrant expression of miR-132 in cardiac cells is causally associated with cardiac remodeling and HF progression.
  Arms: CDR132L 4.52 mg
Drug: Placebo — Placebo to CDR132L
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study including approximately 130 randomized HF patients with heart failure with mildly reduced or preserved ejection fraction (LVEF ≥45%), to assess efficacy and safety of CDR132L on reverse remodeling. In this study, patients with HFpEF (EF ≥50%) or HFmrEF (LVEF 45-49%) will be included.

ELIGIBILITY:
Main Inclusion Criteria:

1. Provision of signed informed consent prior to any study-specific procedures.
2. Male or female of non-childbearing potential patients age ≥40 and <85 years.
3. Documented diagnosis of symptomatic heart failure (NYHA class II-IV) at enrollment, and a medical history of typical symptoms/signs of heart failure ≥6 weeks before enrollment with at least intermittent need for diuretic treatment.
4. Ejection fraction ≥ 45% (determined by echocardiography at site laboratory)
5. Increased intraventricular wall thickness (≥11 mm for female and ≥12 mm for male patients by echocardiography at site laboratory)
6. NT-proBNP > 300 pg/ml (sinus rhythm); >900 pg/ml (atrial fibrillation at time of screening/inclusion or documented with the last 6 months)
7. BMI between 22 kg/m² and 45 kg/m².

Main Exclusion Criteria:

1. Hemoglobin A1C (A1C) ≥10.5%
2. eGFR <35 mL/min/1.73m²
3. Systolic blood pressure (BP) <90 mmHg on 2 consecutive measurements at 5-minute intervals, at Screening.
4. Systolic BP≥180 mmHg on 2 consecutive measurements at 5-minute intervals, at Screening.
5. Planned coronary revascularization, ablation of atrial flutter/fibrillation and valve repair/replacement.
6. Stroke or transient ischemic attack (TIA) within 12 weeks prior to enrolment.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass | 6 months
  Left ventricular mass measured by cardiac magnetic resonance imaging (indexed to the height in meters raised to the power of 2)
Left atrial maximum volume | 6 months
  Left atrial maximum volume (measured by cardiac magnetic resonance imaging in end systole(indexed to the height in meters raised to the power of 2))
Total cardiac extracellular volume | 6 months
  Total cardiac extracellular volume (mL) measured by cardiac magnetic resonance imaging
Left atrial strain | 6 months
  Left atrial strain measured by cardiac magnetic resonance imaging
Maximum left ventricular wall thickness | 6 months
  Maximum left ventricular wall thickness measured by cardiac magnetic resonance imaging
Age-adjusted e' velocity | 6 months
  Age-adjusted e' velocity measured by doppler echocardiography. With e´velocity being the maximal velocity of mitral annular motion (E-wave).
Global longitudinal strain | 6 months
  Global longitudinal strain measured by echocardiography
E/e' | 6 months
  E/e' measured by doppler echocardiography to evaluate the LV filling pressure.
Concentration of N-terminal pro B-type natriuretic peptide | 6 months
  Concentration measured as biomarker from blood samples.
Concentration of high-sensitivity cardiac troponin T | 6 months
  Concentration measured as biomarker from blood samples.

IPD SHARING:
Plan to Share IPD: No